CLINICAL TRIAL: NCT05419700
Title: Patient Characteristics, Treatment Patterns and Outcomes of Advanced Non-small Cell Lung Cancer Patients With EGFR Exon 20 Insertion Mutations: A Non-interventional Retrospective Medical Chart Review in Spain
Brief Title: A Spanish Medical Record Review of Clinical Characteristics and Outcomes in Non-small Cell Lung Cancer Participants With EGFR Exon 20 Insertion
Acronym: ermEX-20
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-788-5009
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Advanced NSCLC With EGFR Exon 20 Insertions Mutations: All participants diagnosed with advanced NSCLC with Epidermal growth factor receptor EGFR exon 20 insertion mutations will be enrolled in this study. All study data will be collected retrospectively from participants medical records via medical chart review.

SUMMARY:
The main aim is to evaluate sociodemographic and clinical characteristics of advanced Non-Small Cell Lung Cancer (NSCLC) in adults participants with epidermal growth factor receptor (EGFR) exon 20 insertions mutations during the 5 years before data extraction date (from 1-Jan-2017 to 1-Jan-2022).

Participants will not receive any drug. This study will only collect the data from the medical records via chart review.

DETAILED DESCRIPTION:
This is an observational, non-interventional, retrospective study in participants with NSCLC with EGFR exon 20 insertions mutations. This study will assess the sociodemographic and clinical characteristics of advanced NSCLC participants.

The study will enroll approximately 60 participants. Participants who were evaluated and treated at the participating sites between 01 January 2017 and 30 September 2021 will be included. The data will be collected from the medical record of participants via medical chart review. All the participants will be assigned to a single observational cohort:

• Participants With Advanced NSCLC with EGFR Exon 20 Insertions Mutations

This multi-center trial will be conducted in Spain. The overall duration of the study will be approximately 27 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a pathologically and/or cytologically confirmed diagnosis of advanced stage NSCLC (International Classification of Disease, 10th revision [ICD-10] C34.x), either primary, advanced or after relapse of initial non-metastatic disease, evaluated and treated during the last five years prior data extraction date from 1-Jan-2017 to 1-Jan-2022.
2. Participants with detection of an EGFR exon 20 insertion mutation, at any point.
3. Has documentation available for at least 2 visits since the initiation of the last treatment within the last five years (1-January-2017 to 1-January-2022).

Exclusion Criteria:

1. Participants do not meet any of the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with advanced NSCLC with EGFR exon 20 insertion and who received treatment during the last 5 years at participating sites will be included in this study.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Based on Type of EGFR Mutation | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  Percentage of participants will be reported based on type of EGFR mutation and its variant: EGFR exon 20 insertion or compound mutations.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  ORR is defined as the percentage of participants on a given treatment that have at least one partial remission (PR)/complete remission (CR) assessment determination within 3 months after initiation of treatment. CR: defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. ORR will be assessed by Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).
Progression-free Survival (PFS) | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  PFS is defined as the time from treatment start until disease progression (PD) or death. PD: defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of longest diameter recorded since the treatment started or the appearance of one or more new lesions. PFS will be assessed by RECIST 1.1.
Disease Control Rate (DCR) | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  DCR is defined as the percentage of participants on a given treatment that have at least one PR/CR/stable disease (SD) and no PD assessment determination within 3 months after treatment start. CR: defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: defined as at least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions. SD: defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD: defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of longest diameter recorded since the treatment started or the appearance of one or more new lesions. DCR will be assessed by RECIST 1.1.
Time-to-treatment Failure (TTF) | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  TTF is defined as the time from treatment start until treatment discontinuation due to any reason including toxicity, PD, or death. PD: defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of longest diameter recorded since the treatment started or the appearance of one or more new lesions. TTF will be assessed by RECIST 1.1.
Overall Survival (OS) | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  OS is defined as the time from treatment start until death from any cause or the last follow-up. OS will be assessed by RECIST 1.1.
Health Care Resources Utilization | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  Health care resources utilization including information related with direct costs (hospitalizations, tests, computed tomography [CT], positron emission tomography [PET], magnetic resonance imaging [MRI]) will be reported.
Percentage of Participants With Grade 3 or Higher Treatment-related Adverse Events (AEs) | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  Treatment-related grade 3 or higher AE will be reported. Treatment-related AE grades will be evaluated as per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Number of Participants who Experience at Least one Treatment-related AE | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  Participants with at least one treatment-related AE will be reported. An AE is defined as any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, a new disease or worsening in severity or frequency of a concomitant disease, temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.
Percentage of Participants who Experience at Least one AEs Leading to Treatment Discontinuation | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
Percentage of Participants Based on Method of Molecular Testing for EGFR Mutation | From the treatment start date till the data extraction date (1-Jan-2017 to 1-Jan-2022)
  Participants will be reported based on the method of molecular testing to analyze EGFR mutations (for example, polymerase chain reaction [PCR], PCR-reverse transcription [RT], Next-generation sequencing [NGS]).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (15):
- Spain (15):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - ICO Badalona. Hospital Universitario Germans Trias i Pujol, Badalona, Catalonia
  - Hospital Clinicde Barcelona, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - ICO Girona. Hospital Universitario Dr. Josep Trueta, Girona, Catalonia
  - Complejo Hospitalario Universitario A Coruna (CHUAC), A Coruña, Galicia
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, Galicia
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid, Madrid
  - Hospital Universitario de Navarra (HUN), Pamplona, Navarre
  - Hospital General Universitario de Alicante, Alicante, Valencia
  - Hospital Universitari i Politecnic la Fe, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5fc45a6963bf47ce?idFilter=%5B%22TAK-788-5009%22%5D